CLINICAL TRIAL: NCT02636153
Title: the Effects of Different Dietary Phosphorus Intake on the Circadian Pattern of Serum Phosphate in Normal Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Chen Jing, Professor, Huashan Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: HuashanH
Record Dates: First submitted 2015-12-09; First posted 2015-12-21 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Healthy
Keywords: phosphorus,dietary; circadian rhythm; phosphorus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Normal Phosphorus Diet (Experimental): Diet containing 1500mg of phosphorus per day
  Interventions: Other: normal diet
- Restricted Phosphorus Diet (Experimental): Diet containing 500mg of phosphorus per day
  Interventions: Other: restricted phosphate diet

INTERVENTIONS:
Other: normal diet — Diet containing 1500mg of phosphorus
  Arms: Normal Phosphorus Diet
Other: restricted phosphate diet — Diet containing 500mg of phosphorus
  Arms: Restricted Phosphorus Diet

SUMMARY:
The purpose of this study is to investigate the effects of normal diet and low-phosphate diet on the level and the circadian pattern of serum phosphate concentration in normal subjects and to explore the underlying mechanisms.

DETAILED DESCRIPTION:
Emerging evidence show that serum phosphate concentrations are not only associated with cardiovascular and all-cause mortality in chronic kidney disease (CKD) patients, but also associated with the mortality in community population (without history of CKD or cardiovascular disease). The rise of serum phosphate will lead to the elevation of serum plasma fibroblast growth factor 23 (FGF23) and parathyroid hormone (PTH) in healthy people, contributing to bone disorders and left ventricle thickening. Therefore, maintaining normal serum phosphate and reducing postprandial fluctuation of serum phosphate are essential for CKD patients as well as healthy people.

As for serum phosphate modulation by diet, most evidence was focused on CKD patients, less focused on healthy people. An American study in 1980s indicated that phosphorus intake was significantly related with the level of 24-h serum phosphate and the circadian pattern of serum phosphate. However, this study failed to explore the underlying mechanisms and the diet in America is different from that in China. Nowadays, normal diet in China is inclined to having more calories and protein, which warrants high diet phosphorus intake, may contributing to huge fluctuation of serum phosphate and thus elevating the incidence and mortality of cardiovascular disease. Therefore, what is the level and circadian pattern of serum phosphate concentrations in normal subjects under our native normal diet in China? Is restricted phosphate diet able to alter the level and circadian pattern of serum phosphate? These questions are what the investigator sare eager to answer.

Accumulating evidence suggest that gastrointestinal tract has a vital effect in phosphate modulation. Berndt etc. suggested that in rat, epidermal cells of duodenum and jejunum could sense the gastrointestinal tract phosphate load, rapidly activating the type IIa Na/Pi-cotransporter in the renal tubule cells, leading to the increase of urinary phosphate, without any changes of serum FGF23, PTH and phosphate concentrations. So the author proposed that there had a gastro intestine-kidney axis in phosphate modulation. However, whether this axis exists in human body remains unclear.

Therefore, the investigators plan to conduct a crossover clinical study to evaluate the level and circadian pattern of serum phosphate concentrations modulated by native normal diet and restricted phosphate diet and then to explore the underlying mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18-45 years
* Healthy volunteers: no history of chronic diseases; no active symptoms or physical signs; negative results of electrocardiogram and chest X-ray; biochemical indicators of regular medical examination are within 95%-105% of normal range
* Willingness to sign the consent form approved by an Institutional Review Board and comply with the study protocol
* Body mass index ranged within 18.5-24 kg/m2

Exclusion Criteria:

* Current history of drug or alcohol abuse as assessed by the principal Investigator
* Subject has blood donations or blood loss more than 300ml within three months
* Allergic to more than two foods or drugs
* Subject has psycho-disability or body disability
* Subject has a condition that in the judgment of the Principal Investigator could potentially pose a health risk to the patient while involved in the study
* Subject has participated in the other clinical trials at the same time

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2016-05; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Circadian rhythm of serum phosphorus concentration | 24 hour

SECONDARY OUTCOMES:
Circadian rhythm of plasma fibroblast growth factor 23 (FGF23) | 24 hour
Circadian rhythm of parathyroid hormone (PTH) | 24 hour
Circadian rhythm of 1, 25-dihydroxyvitamin D (1,25(OH)2D3) | 24 hour
Circadian rhythm of matrix extracellular phosphoglycoprotein (MEPE) | 24 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan hospital, Shanghai Medical College, Fudan University, Shanghai, Shanghai Municipality, China